CLINICAL TRIAL: NCT00793195
Title: Can SMOFlipid®, A Composite Parenteral Nutrition Lipid Emulsion, Prevent Progression Of Parenteral Nutrition Associated Liver Disease In Infants? A Pilot Double Blind Randomized Controlled Trial
Brief Title: Can SMOFlipid®, A Composite Parenteral Nutrition Lipid Emulsion, Prevent Progression Of Parenteral Nutrition Associated Liver Disease In Infants?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Dr. Paul Wales, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000012566
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Short Bowel Syndrome; Intestinal Failure; Gastrointestinal Motility Disorder; Mucosal Enteropathy
Keywords: Neonates; Short Bowel Syndrome; Intestinal Failure; Liver Failure; Parenteral Nutrition; Intralipid; SMOF
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure; Liver Failure; Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1) Intralipid (Active Comparator): Fat Emulsions for Intravenous Nutrition
  Interventions: Drug: Intralipid 20%
- 2) SMOFlipid (Experimental): Fat Emulsions for Intravenous Nutrition
  Interventions: Drug: SMOFlipid 20%

INTERVENTIONS:
Drug: Intralipid 20% — Dosing will be formulated according to a Nomogram for Parenteral Nutrition (PN) composition, which takes into account the percentage of the subject's caloric intake consumed parenterally. PN solution will be infused continuously over 12-24 hours by infusion pump, and the duration each day will depend on the enteral tolerance of the child. PN shall not be discontinued, unless the patient is taking 95% of calories enterally with good growth as evidence by appropriate weight gain. Subjects will receive the trial lipid for a total duration of 12 weeks or if they develop a serum conjugated bilirubin (sustained for 7 days) of 100 umol/l (6mg/dl) or full enteral tolerance prior to this end-point. Once the trial lipid is discontinued, in the event that PN is continued, subjects will return to the standard lipid preparation. A final follow-up data-point will be collected 4 weeks after the trial lipid is stopped.
  Arms: 1) Intralipid
Drug: SMOFlipid 20% — Dosing will be formulated according to a Nomogram for Parenteral Nutrition (PN) composition, which takes into account the percentage of the subject's caloric intake consumed parenterally. PN solution will be infused continuously over 12-24 hours by infusion pump, and the duration each day will depend on the enteral tolerance of the child. PN shall not be discontinued, unless the patient is taking 95% of calories enterally with good growth as evidence by appropriate weight gain. Subjects will receive the trial lipid for a total duration of 12 weeks or if they develop a serum conjugated bilirubin (sustained for 7 days) of 100 umol/l (6mg/dl) or full enteral tolerance prior to this end-point. Once the trial lipid is discontinued, in the event that PN is continued, subjects will return to the standard lipid preparation. A final follow-up data-point will be collected 4 weeks after the trial lipid is stopped.
  Arms: 2) SMOFlipid

SUMMARY:
The aim of this study is to determine the feasibility of conducting a trial to examine the efficacy of an ω3FA (Omega-3 fatty acid) containing balanced lipid emulsion in the prevention of progression of PNALD in infants with Intestinal Failure/Short Bowel Syndrome (SBS) and early liver dysfunction.

DETAILED DESCRIPTION:
Parenteral nutrition (PN) associated liver disease (PNALD), remains the primary cause of morbidity and mortality in infants with Short Bowel Syndrome (SBS) and intestinal failure. Although, the etiology is likely multi-factorial, lipids within parenteral nutrition solution have been implicated in its development. The standard lipid used in PN is typically, a soy based lipid (eg: Intralipid® - Fresenius Kabi) that primarily contains omega-6 fatty acids (ω6FAs). Animal and human studies have suggested that addition of omega-3 fatty acids (ω3FAs) to parenteral nutrition may decrease the incidence of hepatic injury, as well as have beneficial immunologic effects. SMOFlipid® (Fresenius Kabi) is a composite lipid emulsion, which contains polyunsaturated ω3 and ω6FAs, monounsaturated FAs, as well as medium chain FAs as integral constituents. All components (Soy-bean oil, medium chain triglycerides, olive oil, fish oil) have been used in humans, and the drug is approved for use in children in Europe. Based on its composition, we believe that this lipid preparation has the potential to prevent progression of liver disease in infants with SBS who are demonstrating evidence of liver dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. ≤ 24 months of age at enrollment
2. Evidence of early hepatic dysfunction

   * Serum conjugated bilirubin ≥ 17 umol/L on 2 consecutive readings 7 days apart

     * No evidence of sepsis

       * Normal Temperature (T between 35.5C and 38.0C)
       * Normal leukocyte count
       * Normal platelet count
       * No systemic septic symptoms
     * No prior administration of Omegaven
3. ≥ 40% of total calories administered by PN
4. Meet one of the following diagnostic categories

   * Short Bowel Syndrome

     * Abdominal surgical procedure including gastroschisis closure by any means and percutaneous drainage procedures within the past 6 months and has been receiving PN since surgery
   * Intestinal Failure

     * One of the following diagnoses for which the child is dependent on PN

       * Gastrointestinal Motility Disorder
       * Mucosal Enteropathy
5. Expectation of the treating physician that the patient will require PN for at least 3 weeks following enrollment.
6. Parents willing to participate including randomization

Exclusion Criteria:

1. Sepsis or Hemodynamic Instability of any cause.
2. Coagulopathy (Platelets ≤ 150 000, or INR ≥ 1.4)
3. Hypersensitivity to fish-, egg- or soy protein or to any of the active substances or excipients
4. Current enrollment in another clinical trial involving a surgical or pharmacologic intervention
5. Serum conjugated bilirubin > 50 umol/L
6. Hyperlipidaemia (any of)

   * LDL ≥ 4 mmol/L
   * HDL ≥ 2 mmol/L
   * Total cholesterol ≥ 5 mmol/L
   * Triglycerides ≥ 1.5 mmol/L
7. Treatment with intravenous N-Acetylcysteine or Ursodeoxycholic acid
8. Renal insufficiency

   * Creatinine ≥ 80 umol/L
9. Disorders of Fluid Balance (any of)

   * Serum Sodium < 130 mmol/L
   * Serum Sodium > 145 mmol/L
10. Unstable conditions

    * Acute pulmonary edema
    * Decompensated cardiac insufficiency
    * Severe post-traumatic conditions
    * Uncompensated diabetes mellitus
    * Acute myocardial infarction
    * Stroke within 3 months
    * Thromboembolic event within 3 months
    * Metabolic acidosis

      * Serum Bicarbonate < 17 mmol/L

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Mean serum conjugated bilirubin (umol/L) | 12 weeks

SECONDARY OUTCOMES:
Proportion with the development of cholestasis (sustained serum conjugated bilirubin >50 umol/L for greater than 2 weeks in absence of sepsis) | 12 and 16 weeks
Proportion with progression of liver disease (sustained serum conjugated bilirubin >100 umol/L in absence of sepsis) | 12 and 16 weeks
Degree of enteral tolerance (%) | 12 and 16 weeks
Growth parameters | 12 and 16 weeks
Biochemical outcomes shall assess mean levels of "hepatic markers" (AST, ALT, ALP, GGT), coagulation parameters (PT, PTT, INR, platelets), serum lipid levels (triglycerides and cholesterol), serum albumin, and Nephelometry (lipid clearance). | 12 and 16 weeks
Immunologic outcomes shall include assessment of RBC phospholipids composition, C-reactive Protein (CRP) and serum immunologic marker (IL-1b, IL-2R, IL-6, IL-8, IL-10, TNF-α) assessment | 12 and 16 weeks
Feasibility of trial (recruitment, protocol adherence, estimated effect size | 4, 12 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wales, Principal Investigator — The Hospital for Sick Children
Locations (5):
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - Foothills Medical Center, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Hamilton Health Sciences, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Diamond IR, Grant RC, Pencharz PB, de Silva N, Feldman BM, Fitzgerald P, Sigalet D, Dicken B, Turner J, Marchand V, Ling SC, Moore AM, Avitzur Y, Wales PW. Preventing the Progression of Intestinal Failure-Associated Liver Disease in Infants Using a Composite Lipid Emulsion: A Pilot Randomized Controlled Trial of SMOFlipid. JPEN J Parenter Enteral Nutr. 2017 Jul;41(5):866-877. doi: 10.1177/0148607115626921. Epub 2016 Feb 2. PMID 26838529